Date: 9/7/2022

National Clinical Trials #: NCT05219422

Study Title: Improving the Implementation of Evidence-based Drug Prevention Programs in Schools

## PARENT/LEGAL GUARDIAN CONSENT FORM FOR CHILD'S SURVEY PARTICIPATION Project ALERT

| <b>PRINT</b> r | name of your child: | | | | |
|---|---|---|---|---|---|
| | • | First Name | Middle Name | Last N | lame |
| | ad (or someone has rea<br>ion Letter which explair | • | | = | T Survey |
| lease m<br>Agree<br>Refuse | nark "Agree" or "Refuse<br>I agree to allow my chi<br>measure change in att<br>I refuse to allow my ch | ld to complete t<br>itudes and beha | viors. | | · |
| ~~~~ | SIGNAT | URE OF PARENT | OR LEGAL GUAF | RDIAN | |
| Today's | date:/ | / | | | |
| Are you | the child's: | Parent | Legal Guardian | | |
| Parent/ | Legal Guardian's Addre | ss: | | | |
| City, State: | | | Zip: | | |
| Parent/ | Guardian's Telephone N | lumber: | | | |
| Parent/ | Guardian's Email Addre | ss: | | | |
| Print NA | AME of parent or legal g | uardian: | | | |
| | | | First | Middle | Last |
| | SIG | NATURE of pare | nt or legal guardia | an | |

Please return to RAND in the included pre-paid envelope, or to your child's teacher.

RAND Corporation
ATTN: Survey Research Group - Data Reduction
Project ALERT
1776 Main Street
Santa Monica, CA 90401